CLINICAL TRIAL: NCT00577187
Title: Placement of Coronary Sinus/Left Ventricular Leads With EnSite NavX Guidance
Brief Title: Placement of CS/LV Pacing Leads With EnSite NavX Guidance
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0712.0
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EnSite NavX-Guided CRT implant — LV lead placement during CRT implant using EnSite NavX

SUMMARY:
This study utilizes the 3D mapping capabilities of the EnSite NavX mapping system to help guide the placement of the left ventricular lead during cardiovascular resynchronization therapy implant procedures with the goal of reducing fluoroscopic exposure and procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Patients schedule to undergo CRT implant (per established guidelines)

Exclusion Criteria:

* Standard exclusions to CRT implant procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Fluoroscopy and procedure time | Procedural

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Erickson, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States